CLINICAL TRIAL: NCT02405819
Title: Patient and Provider Initiated Survivorship Care Planning: a Randomized Pilot Study
Brief Title: Patient and Provider Initiated Survivorship Care Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genentech, Inc. (Industry); WellPoint, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: J14178; IRB00057614 (Other: JHMIRB)
Record Dates: First submitted 2015-03-13; First posted 2015-04-01 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2015-11

CONDITIONS: Cancer
Keywords: Cancer; Oncology; Survivorship; Care; Plan
MeSH Terms: conditions — Neoplasms; Neuroaxonal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Directed (Other): We will collect baseline data, including sociodemographic information for the patients and an assessment of each patient's baseline supportive care needs and knowledge about survivorship care. Sociodemographic information will be self completed. All other data collection will be interviewer administered. The instruments used at baseline and follow-up are adapted from previously published surveys (Hodgkinson et al, 2007; Sprague et al, 2013; Griggs et al). The research team will direct patients to their assigned condition by providing a hand-out directing them to the planning tool. After 2 months, we will re-contact all randomized patients to determine whether the survivorship care planning occurred as intended.
  Interventions: Other: 'My Care Plan'
- Clinician Directed (Other): We will collect baseline data, including sociodemographic information for the patients and an assessment of each patient's baseline supportive care needs and knowledge about survivorship care. Sociodemographic information will be self completed. All other data collection will be interviewer administered. The instruments used at baseline and follow-up are adapted from previously published surveys (Hodgkinson et al, 2007; Sprague et al, 2013; Griggs et al). The provider will be provided a hand-out with their patient's assigned condition and is responsible for implementing the survivorship care plan process. After 2 months, we will re-contact all randomized patients to determine whether the survivorship care planning occurred as intended.
  Interventions: Other: 'Survivorship Care Plan Builder'

INTERVENTIONS:
Other: 'My Care Plan' — 'My Care Plan' is a patient-initiated survivorship care planning tool.
  Arms: Patient Directed
Other: 'Survivorship Care Plan Builder' — 'Survivorship Care Plan Builder' is a provider-initiated survivorship care planning tool.
  Arms: Clinician Directed

SUMMARY:
Objective: to describe and compare the implementation of two cancer survivorship care tools: (1) 'My Care Plan': a patient-initiated tool and (2) 'Survivorship Care Plan Builder': a provider-initiated tool. The results of this study will be used to (1) provide an initial assessment of the two survivorship care planning tools and (2) inform the design and conduct of a larger study.

DETAILED DESCRIPTION:
Background/Rationale: In a 2005 report 'From Cancer Patient to Cancer Survivor: Lost in Transition', the Institute of Medicine recommended that cancer patients completing treatment receive a summary of the care received and a plan outlining follow-up care needs. Taken together these materials are referred to as a 'Survivorship Care Plan', or SCPs. Based on this recommendation from the IOM, a number of organizations developed survivorship care plan templates. Two of these templates, 'Survivorship Care Plan Builder' and 'My Care Plan,' were developed by Journey Forward, a collaboration among the National Coalition for Cancer Survivorship, UCLA Cancer Survivorship Center, Oncology Nursing Society, WellPoint, Inc., and Genentech (http://journeyforward.org/). These tools are available free of charge to those wishing to use them. As the time and effort required to complete SCP documents have been found to be barriers to implementation, this study aims to explore the use of these two tools.

Research Questions:

1. What processes are undertaken to implement survivorship care planning?

   * How do these processes differ between the patient-initiated My Care Plan and provider-initiated Survivorship Care Plan Builder?
2. What is the feasibility of implementing survivorship care planning?

   * Does the feasibility differ between the patient-initiated My Care Plan and provider-initiated Survivorship Care Plan Builder?
3. What is the value of survivorship care planning to both patients and providers?

   * Does the value differ between the patient-initiated My Care Plan and provider-initiated Survivorship Care Plan Builder?

Study Design: This is a pilot randomized study. Cancer patients completing acute treatment with a participating provider will be randomized to either the patient-initiated My Care Plan tool or provider-initiated Survivorship Care Plan Builder. The investigators will describe and compare how each tool is implemented in practice, the feasibility of completing each tool, and the value of the tools to patients and providers. The study will use quantitative and qualitative measures of implementation, feasibility, and value.

ELIGIBILITY:
Inclusion Criteria:

1. Have you diagnosed with non-metastatic (i.e., stages I - III) cancer (non-melanoma skin cancer)
2. Have you completed acute treatment with intent to cure within the past 2 months (ongoing long-term maintenance therapy such as adjuvant hormonal therapy is allowed)
3. What clinician primarily managed your cancer treatment? (must be a participating Sibley or Suburban clinician)

Exclusion Criteria:

1. Do you show any evidence of disease?

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Patient in receipt of a complete survivorship care plan | 16 weeks
  As this study explores the feasibility of the survivorship care planning process, the primary outcome measure is whether or not the patient receives a complete survivorship care plan.

SECONDARY OUTCOMES:
Change in score for the CaSUN (Cancer Survivors' Unmet Needs) assessment tool | 16 weeks
  The change in score on the CaSUN tool will be used to asses the value of survivorship care planning.
Change in score on the PLANS (Preparing for Life as a New Survivor) assessment tool | 16 weeks
  The change in score on the PLANS tool will be used to asses the value of survivorship care planning.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Smith, Ph.D., Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland

REFERENCES:
- [Background] Griggs, J. et al. PLANS ("Preparing for Life as a New Survivor")
- [Background] Hodgkinson K, Butow P, Hunt GE, Pendlebury S, Hobbs KM, Lo SK, Wain G. The development and evaluation of a measure to assess cancer survivors' unmet supportive care needs: the CaSUN (Cancer Survivors' Unmet Needs measure). Psychooncology. 2007 Sep;16(9):796-804. doi: 10.1002/pon.1137. PMID 17177268
- [Background] Sprague BL, Dittus KL, Pace CM, Dulko D, Pollack LA, Hawkins NA, Geller BM. Patient satisfaction with breast and colorectal cancer survivorship care plans. Clin J Oncol Nurs. 2013 Jun;17(3):266-72. doi: 10.1188/13.CJON.17-03AP. PMID 23722604
- [Derived] Smith KC, Tolbert E, Hannum SM, Radhakrishnan A, Zorn K, Blackford A, Greco S, Smith K, Snyder CF. Comparing Web-Based Provider-Initiated and Patient-Initiated Survivorship Care Planning for Cancer Patients: A Randomized Controlled Trial. JMIR Cancer. 2016 Aug 30;2(2):e12. doi: 10.2196/cancer.5947. PMID 28410187
- See also: Journey Forward is a cancer survivorship program for healthcare providers and patients who have finished active treatment. — http://www.journeyforward.org/